CLINICAL TRIAL: NCT06303167
Title: MATCH Treatment Subprotocol E: Osimertinib (AZD9291) in Patients With Tumors Having EGFR T790M Mutations or Rare Activating Mutations of EGFR
Brief Title: Testing AZD9291 as Potentially Targeted Treatment in Cancers With EGFR Genetic Changes (MATCH-Subprotocol E)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01150; NCI-2024-01150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-E (Other: ECOG-ACRIN Cancer Research Group); EAY131-E (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-03-08; First posted 2024-03-12 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; osimertinib; X-Rays

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (osimertinib) (Experimental): Patients receive osimertinib (AZD9291) PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, ECHO or MUGA during screening, and biopsy and collection of blood samples on trial and at end of treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Osimertinib; Procedure: Radiologic Examination

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
Procedure: Radiologic Examination — Undergo radiologic evaluation
  Other Names: Radiologic Evaluation; Radiologic Exam

SUMMARY:
This phase II MATCH treatment trial evaluates the effectiveness of osimertinib (AZD9291) in treating patients with cancer that has certain genetic changes called EGFR mutations. Osimertinib is in a class of medications called kinase inhibitors. It works by blocking the action of mutant forms of the EGFR protein, which play a key role in tumor cell growth. Osimertinib may cause tumor cell death and inhibit tumor growth in EGFR-overexpressing tumor cells, thereby stopping or slowing the spread of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive osimertinib (AZD9291) orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening, and biopsy and collection of blood samples on trial and at end of treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patient must fulfill all eligibility criteria outlined in MATCH Master Protocol at the time of registration to treatment step (step 1, 3, 5, 7)
* Patients must have either of the below, or another aberration, as determined via the MATCH Master Protocol:

  * Any malignancy except non-small cell lung cancer (NSCLC) with EGFR T790M identified in their tumor, with or without an activating mutation OR
  * Any malignancy harboring any of the following mutations: EGFR G719A, G719C, G719D, G719S EGFR L861Q, S786I or an EGFR exon 19 in frame insertion mutation
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block, and second-degree heart block
* Patients must have an ECHO or a nuclear study (MUGA or first pass) within 4 weeks prior to registration and must not have a left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients must not have known hypersensitivity to osimertinib (AZD9291) or compounds of similar chemical or biologic composition or any of the inactive excipients of the tablets
* Patient must not have received osimertinib (AZD9291), WZ4002, CO-1686, HM61713, EGF816 or ASP8273 previously
* Patients known to harbor germline EGFR T790M mutations are excluded from the study. Prospective testing for germline mutations is not required
* Patients must not have a history of interstitial lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, radiation pneumonitis requiring steroids, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients must not currently be receiving treatment with potent CYP3A4 inducters or medications "known to prolong" the QT interval. Drugs that "may possibly prolong" the QT interval, are permitted if the patient has been stable on therapy for the period indicated for the specific medication
* Patients must agree to not donate sperm from the start of protocol treatment until at least 4 months after the last dose of protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V Sequist, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol E was activated on August 12, 2015. Nineteen patients were enrolled between January 2016 and November 2021. Three patients were enrolled on the basis of the results from the NCI-MATCH assay and 16 on the basis of the outside assay results.
Pre-assignment Details: Patients with an EGFR T790M mutation in any histology except lung cancer and patients with a rare activating mutation (EGFR G719A, G719C, G719D, G719S, L861Q, S786I, or an exon 19 in frame insertion mutations) in any histology were offered participation in this subprotocol. The mutation status was determined by a CLIA-approved assay performed in an NCI-MATCH approved laboratory for 16 patients in this arm, these cases had to be confirmed to be used in primary analysis.
Groups:
- Treatment (Osimertinib): Patients receive osimertinib (AZD9291) 80 mg PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo radiologic evaluation throughout the trial, ECHO or MUGA during screening, and biopsy and collection of blood samples on trial and at end of treatment.
Period: Overall Study
Arm/Group | Treatment (Osimertinib)
Started | 19
Started Protocol Therapy | 17
Eligible and Treated | 16
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 13
Completed | 0
Not Completed | 19
Not completed — Ineligible | 1
Not completed — Never start protocol therapy | 2
Not completed — Disease progression | 16

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 13
percentage of participants | 15.4 [2.8 to 41]

2. Secondary Outcome: 6-month Progression-Free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 13
percentage of participants | 16.7 [0 to 34.4]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 13
months | 2.7 [1.74 to 4.04]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Seventeen patients were included in the toxicity analysis (excluding two who did not receive treatment).
Arm/Group | Treatment (Osimertinib)
All-Cause Mortality (participants affected / at risk) | 14/19
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Osimertinib) (N=17)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Osimertinib) (N=17)
Anemia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Fatigue (General disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Paronychia (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT06303167/Prot_000.pdf